CLINICAL TRIAL: NCT01489085
Title: Etude Clinique Observationnelle, Prospective, Ouverte, Monocentrique Sur l'Utilisation d'un Mode Ventilatoire entièrement automatisé Chez Les Patients de réanimation de l'Intubation Jusqu'au Sevrage.
Brief Title: Observational Study Evaluating the Use of Intellivent® for Patients With Respiratory Distress Syndrome
Acronym: intellivent
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Other Study IDs: S1FRTOU-3
Record Dates: First submitted 2011-12-06; First posted 2011-12-09 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2010-11

CONDITIONS: Respiratory Distress Syndrome
Keywords: ventilation; automated
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Rational: Intellivent is a ventilation mode completely automated which controls ventilation and oxygenation parameters. Safety and performance of IntelliVent has still been demonstrated in post operative heart surgery for patient with a controlled ventilation on short period (2 to 4 hours). This feasibility study evaluate the use of Intellivent for Intensive care unit patients from intubation to coming off.

Primary objective : Compare parameters which have been selected by automated mod (Intellivent) to those selected by clinical practitioner in a conventional mode

Secondary objectives: Record oxygenation , gaseous interchange and ventilation parameters. Record complications, number of manual adjustments and prognostic signs.

Methodology: Patients in the intensive care unit who need invasive ventilation. They will be included after a detailed information (information note). Oxygenation and ventilation parameters will be recorded 2 times by day from intubation to coming off. The investigator in charge will determine daily at the bedside of the patient the adjustments he should make in a conventional mode. These adjustments will be compared to the IntelliVent automated adjustments.

Experimental study, observational, prospective, comparative, opened, monocentric in an intensive care unit.

Number of patients: 100

ELIGIBILITY:
Inclusion Criteria:

* Patient which needs an invasive ventilation
* Intubation < 24 hours
* Age ≥ 18 years

Exclusion Criteria:

* Patient which has withdrawal standard in line with the unit coming off procedure (all criteria must be present)
* temperature ≤ 38,5°C
* No pressor drug
* No sedation,
* Motor response to order,
* Cough during bronchoaspiration
* %VM ≤ 130%, FiO2 ≤ 50%, PEEP ≤ 5 cmH2O, Pinsp ≤ 25 cmH2O.
* Patient with non invasive ventilation .
* Dysfunctions of the ventilatory command (ex Cheyne-Stokes).
* Broncho pleural fistula.
* Brain dead status.
* Pregnant woman.
* Adult under guardianship.
* Person deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive care Unit intubated Patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
oxygenation , gaseous interchange and ventilation parameters | Participants are followed until they no longer need ventilation up to 10 days
  Record oxygenation , gaseous interchange and ventilation parameters

CONTACTS AND LOCATIONS:
Overall Officials: jean-michel arnal, ph, Principal Investigator — Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer
Locations (1):
- Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer, Toulon, France

REFERENCES:
- [Background] Arnal JM, Wysocki M, Nafati C, Donati S, Granier I, Corno G, Durand-Gasselin J. Automatic selection of breathing pattern using adaptive support ventilation. Intensive Care Med. 2008 Jan;34(1):75-81. doi: 10.1007/s00134-007-0847-0. Epub 2007 Sep 11. PMID 17846747
- [Derived] Arnal JM, Garnero A, Novonti D, Demory D, Ducros L, Berric A, Donati S, Corno G, Jaber S, Durand-Gasselin J. Feasibility study on full closed-loop control ventilation (IntelliVent-ASV) in ICU patients with acute respiratory failure: a prospective observational comparative study. Crit Care. 2013 Sep 11;17(5):R196. doi: 10.1186/cc12890. PMID 24025234